CLINICAL TRIAL: NCT04260113
Title: The Effectivity and Toxicity of Apatinib for Unresectable Advanced Chondrosarcoma: a Multicentric Retrospective Study
Brief Title: Apatinib for Inoperable Advanced Chondrosarcoma
Acronym: AIAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSSG-06
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Efficacy; Toxicity, Drug
Keywords: chondrosarcoma; apatinib; inoperable; toxicity; prognosis
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Chondrosarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Arm (Experimental)
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib orally 500mg once daily half an hour after meal

SUMMARY:
Anti-angiogenesis Tyrosine kinase inhibitors (TKIs) have been proved to show promising effects on prolonging progression-free survival (PFS) for advanced chondrosarcoma after failure of standard multimodal Therapy. Methylsulfonic apatinib is one of those TKIs which specifically inhibits VEGFR-2. This study summarizes the experience of two Peking University affiliated hospitals in off-label use of apatinib in the treatment of extensively pre-treated chondrosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed high-grade sarcoma;
* 2) initial treatment in the orthopedic oncology departments of the two affiliated hospitals of Peking University;
* 3) tumors not amenable to curative treatment or inclusion in clinical trials;
* 4) unresectable local advanced lesions or multiple metastatic lesions that could not be cured by local therapy;
* 5) measurable lesions according to Response Evaluation Criteria for Solid Tumors (RECIST1.1) ;
* 6) Eastern Cooperative Oncology Group performance status 0 or 1;
* 7) acceptable hematologic, hepatic, and renal function.

Exclusion Criteria:

* had central nervous system metastasis;
* had other kinds of malignant tumors at the same time; had cardiac insufficiency or arrhythmia;
* had uncontrolled complications such as diabetes mellitus, coagulation disorders, urine protein ≥ ++ and so on;
* had pleural or peritoneal effusion that needs to be handled by surgical treatment;
* combined with other infections or wounds;
* pregnant or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  from initial treatment to date of recorded progression or death or last follow-up

SECONDARY OUTCOMES:
overall survival | 5 years
  from initial treatment to death or last follow-up
objective response rate | 6 months
  CR+PR according to RECIST 1.1
clinical benefit rate | 6 months
  CR+PR+SD according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Musculoskeletal Tumor Center of Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking Univresity Shougang Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie L, Guo W, Wang Y, Yan T, Ji T, Xu J. Apatinib for advanced sarcoma: results from multiple institutions' off-label use in China. BMC Cancer. 2018 Apr 6;18(1):396. doi: 10.1186/s12885-018-4303-z. PMID 29625604
- [Background] Xie L, Xu J, Sun X, Tang X, Yan T, Yang R, Guo W. Apatinib for Advanced Osteosarcoma after Failure of Standard Multimodal Therapy: An Open Label Phase II Clinical Trial. Oncologist. 2019 Jul;24(7):e542-e550. doi: 10.1634/theoncologist.2018-0542. Epub 2018 Dec 17. PMID 30559126
- [Result] Xie L, Xu J, Sun X, Liu K, Li X, He F, Liu X, Gu J, Lv Z, Yang R, Tang X, Yan T, Li D, Yang Y, Dong S, Sun K, Shen D, Guo W. Apatinib for Treatment of Inoperable Metastatic or Locally Advanced Chondrosarcoma: What We Can Learn About the Biological Behavior of Chondrosarcoma from a Two-Center Study. Cancer Manag Res. 2020 May 15;12:3513-3525. doi: 10.2147/CMAR.S253201. eCollection 2020. PMID 32547189